CLINICAL TRIAL: NCT04832828
Title: Sensitivity and Specificity of the Roth Test in Patients With COVID-19 Positive
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal investigator, Universidad Autonoma de Madrid
Other Study IDs: PI-4321
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COVID+ Group: Patients diagnosed with Covid19 positive in last 7 days
  Interventions: Diagnostic Test: Roth´s Test

INTERVENTIONS:
Diagnostic Test: Roth´s Test — Subjets must count from 1 to 30 in their languages, and health professional will count seconds that last in take breath during the count.

SUMMARY:
The presence of the described silent hypoxia in subjects diagnosed with COVID19 highlights the need for valid tools to assess respiratory capacity. The Roth test has been associated with acceptable sensitivity and specificity criteria in patients with previous respiratory pathology; however, its validity in this type of patient has not been proven.

ELIGIBILITY:
Inclusion Criteria:

1. having been diagnosed as COVID-19 positive and with symptoms compatible with Sars-Cov-2 infection in the last 7 days prior to assessment,
2. having an understanding of Spanish,
3. and having no history of respiratory pathology prior to the current infection.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects aged 18 to 90 years were recruited by non-probabilistic convenience sampling in Primary Health Care Centres of the Primary Health Care Management of SERMAS and the Intensive Care Unit of the University Hospital of Gran Canaria Doctor Negrín of the Canary Health Service
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | 12 weeks
  The pulseoximeter percentage value

SECONDARY OUTCOMES:
Roth´s test | 12 weeks
  The level described in the test

CONTACTS AND LOCATIONS:
Locations (1):
- CS Entrevías, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No